CLINICAL TRIAL: NCT06140420
Title: Naltrexone Treatment for Prolonged Grief Disorder: A Proof of Concept Study
Brief Title: Naltrexone for Prolonged Grief Disorder
Acronym: NPGD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding unexpectedly withdrawn
Sponsor: Texas Tech University (Other)
Collaborators: Texas Tech University Health Science Center (Unknown)
Responsible Party: Principal Investigator, Jonathan Singer, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TexasTechU6
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Naltrexone HCl 50 MG Oral Tablet; Placebo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator: Placebo (Placebo Comparator): 24 randomized patients will take placebo daily for 8 weeks.
  Interventions: Drug: Placebo
- Active Comparator: Naltrexone (Active Comparator): 24 randomized patients will take naltrexone daily for 8 weeks
  Interventions: Drug: Naltrexone Oral Product

INTERVENTIONS:
Drug: Naltrexone Oral Product — Generic, oral tablet.
  Arms: Active Comparator: Naltrexone
Drug: Placebo — Oral Placebo
  Arms: Placebo Comparator: Placebo

SUMMARY:
This is a study to see how effective oral naltrexone is as treatment for prolonged grief disorder (PGD). Participants will take their assigned medication for 8 weeks, with monthly visits to assess symptom severity, social connectedness, and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Lives within a reasonable distance from NYPH for convenient clinic visits.
* Can speak, read, and write English proficiently.
* Meet diagnostic criteria for PGD based on the DSM guidelines
* If a female patient, must agree to use a method of contraception and be willing and able to continue contraception during the first 8 weeks of the study while she is taking the study drug. Female patients who are planning to use oral hormonal contraception during this time must have initiated it at least 2 months prior to the baseline visit.
* If a male patient, must agree to use a method of contraception and be willing and able to continue contraception during the first 8 weeks of the study while he is taking the study drug.

Exclusion Criteria:

• Having recently started taking/prescribed medications for any psychiatric illness (e.g.

SSRIs for MDD) within the past 3 months; participants who have been taking this medication for longer than 3 months can be included.

* Having recently started psychotherapy for any psychiatric illness within the past 3 months; participants who have been receiving psychotherapy for longer than 3 months can be included.
* Prior history of recently active (e.g. within the past 3 months) opioid dependence.
* Current prescription, non-prescription, or illicit opioid use, (i.e., acute use within the past 14 days or chronic use within the last 30 days), including opioid antagonists for alcohol or opioid dependence, all opioid analgesics, certain cough and cold remedies (e.g., codeine), and certain anti-diarrheal preparations (e.g., loperamide).
* Possible future use of opioids during the study (e.g. for surgery).
* Current use of leflunomide (Arava), droperidol (Droleptan), diazepam (Valium), thioridazine (Mellaril, Novoridazine, Thioril), or any other clinically relevant medication that has potential to cause liver injury with concurrent use of naltrexone.
* Currently pregnant, lactating, or planning to become pregnant during the study.
* Active hepatitis or liver disease.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels more than one standard deviation (SD) above the upper limit of normal on initial laboratory examination. Screen positive for active suicidal thoughts or behaviors.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Prolonged Grief Disorder symptom severity as assessed by the PGD-12 | Weekly for 12 weeks
  Change in PGD symptom severity will be measured by using Prolonged Grief-13 (PGD-12), a self-rated scale consisting of 12 items. For this study, we have added an additional item inquiring about loneliness to be congruent with DSM-5-TR criteria and SCIP. This 5-point Likert-type of measurement tool evaluates the intensity and severity of the PGD. The validity and reliability of the PGD-12 was tested and validated in previous studies.
Change in Prolonged Grief Disorder severity as assessed by Structured Clinical Interview for PGD | Every 4 weeks for 8 weeks
  The IOS is a self-reported pictorial tool use to measure the subjectively perceived closeness of a relationship. The tool asks respondents to select one of seven pairs of increasingly overlapping circles that best represents their relationship with another, with more overlap signifying a closer relationship. This scale possesses good reliability, with (α = .93) for the entire sample, (α = .87) for family, (α = .92) for friendship, and (α = .95) for romantic relationships. Test-retest reliability shows similar findings, with (α = .83) for the entire sample, (α = .85) for family, (α = .86) for friendship, and (α = .85) for romantic relationships.

SECONDARY OUTCOMES:
Change in strength of subjectively perceived closeness of a social relationship as measured by the Inclusion of the other in the Self (IOS) Scale | Every 4 weeks for 12 weeks
  The IOS is a self-reported pictorial tool use to measure the subjectively perceived closeness of a relationship. The tool asks respondents to select one of seven pairs of increasingly overlapping circles that best represents their relationship with another, with more overlap signifying a closer relationship. This scale possesses good reliability, with (α = .93) for the entire sample, (α = .87) for family, (α = .92) for friendship, and (α = .95) for romantic relationships. Test-retest reliability shows similar findings, with (α = .83) for the entire sample, (α = .85) for family, (α = .86) for friendship, and (α = .85) for romantic relationships.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech Health Science Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gang J, Kocsis J, Avery J, Maciejewski PK, Prigerson HG. Naltrexone treatment for prolonged grief disorder: study protocol for a randomized, triple-blinded, placebo-controlled trial. Trials. 2021 Feb 1;22(1):110. doi: 10.1186/s13063-021-05044-8. PMID 33522931
- [Background] Kakarala SE, Roberts KE, Rogers M, Coats T, Falzarano F, Gang J, Chilov M, Avery J, Maciejewski PK, Lichtenthal WG, Prigerson HG. The neurobiological reward system in Prolonged Grief Disorder (PGD): A systematic review. Psychiatry Res Neuroimaging. 2020 Sep 30;303:111135. doi: 10.1016/j.pscychresns.2020.111135. Epub 2020 Jul 3. PMID 32629197